CLINICAL TRIAL: NCT04125004
Title: Evaluation of Technology-Based Distractions In Pediatric Patients During General Surgery Minor Procedures
Brief Title: Use of Virtual Reality for Pediatric Minor Surgical Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Exploratory pre-study demonstrated participants unwilling to be randomized to control arm.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephanie D. Chao, Assistant Professor of Pediatric Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 52692
Record Dates: First submitted 2019-09-09; First posted 2019-10-14 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Virtual Reality; General Anesthesia
Keywords: virtual reality; pediatric surgery; general anesthesia; distraction technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality (Experimental): Patients will use virtual reality headset during procedure
  Interventions: Device: Samsung Virtual Reality Headset
- general anesthesia (No Intervention): Patients will undergo general anesthesia for their procedure

INTERVENTIONS:
Device: Samsung Virtual Reality Headset — Patients will pick a game or feature from the virtual reality headset to use during their procedure
  Arms: virtual reality

SUMMARY:
This project is looking to use virtual reality for minor general surgery procedures in addition to local anesthesia instead of general anesthesia.

DETAILED DESCRIPTION:
Study population. Patients ages 7-18 undergoing minor surgical procedures at Lucile Packard Children's Hospital will be recruited. Minor surgical procedures include hormone implant placement/removal/exchange, cecostomy tube exchange, incision and drainage of superficial soft tissue abscesses excluding the perineum and buttock, excision of benign masses <2cm on the extremity (e.g. sebaceous cyst, pilomatricoma, lipoma, etc), and foreign body removal from superficial wounds. Exclusion criteria include those with significant cognitive impairment, history of motion sickness, history of seizures, Glasgow Coma Scale (GCS) <15, currently taking anxiety medication or narcotics, facial trauma, clinically unstable or require urgent/emergent intubation, claustrophobia, and visual or auditory impairment. The investigators aim to enroll at least 200 patients into the study.

Intervention. Research coordinators will recruit patients and their families prior to their schedule procedures. Informed consent and assent will be obtained from participants and their caregivers when a patient is a minor. Demographic information will be collected from all participants. Patients will complete pre-procedural survey for pain and anxiety. Parents will complete a survey that documents their perception of their child's anxiety level. Patients will be randomly assigned to a treatment arm.

Patients assigned to the general anesthesia arm will have a child life specialist in the pre-procedural period per hospital routine. Anesthesia will be administered at the discretion of the anesthesiologist. Once the procedure is completed, the patient will recover and be monitored in the post-anesthesia care unit (PACU) per hospital guidelines.

Patients assigned to the virtual reality arm will be instructed on how to use the handheld system. A trained research coordinator or child life specialist will be with the patient during the procedure to help with any issues that may arise. They will document any interfering behaviors during the procedure. After the procedure, the patient will be monitored in the PACU per hospital guidelines.

All patients will complete the post-procedural survey for pain and anxiety. Patients, parents and the surgeon will also complete satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* less than 18 years of age
* parental consent/patient assent
* undergoing minor procedure(s)

Exclusion Criteria:

* participants and patients who do not consent
* have significant cognitive impairment
* have a history of severe motion sickness
* currently have nausea
* history of seizures or currently experiencing seizures
* have visual or auditory impairment
* clinically unstable or require urgent/emergent intervention and/or American Society of Anesthesiologist class 4 or 5
* history of claustrophobia
* Glasgow Coma Scale <15
* currently taking anxiety medication
* currently taking narcotics
* facial trauma

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Completion of procedure | 2 years
  Can the procedure be completed without general anesthesia or procedure sedation. Surgeons will be provided with a self-report survey documenting completion of the procedure. This will be assessed by the surgeon completing the procedure who will answer via questionnaire.

SECONDARY OUTCOMES:
Change in Children's Fear Scale | 2 years
  The Children's Fear Scale (McMurty et al. 2011) is a self-reported scale that uses cartoon depictions of faces to quantify on a 0-4 scale how scared a child is at the given moment
Pain Catastrophizing Scale for Parents | 2 years
  Parents will complete a modified Pain Catastrophizing Scale for Parents (PCS-P) before and after the procedure. This survey identifies the thoughts and feelings of the parent in relation to the pain their child may experience during the procedure. Scores range from 1 (not at all) to 5 (very much).
Change in Faces Pain Scale | 2 years
  The Face Pain Scale (Hicks et. al., 2001) is a self-reported scale that uses cartoon depictions of faces to quantify on a scale 0-10 scale how pain a child is experiencing at a given moment.
Caregiver's satisfaction of procedure | 2 years
  A satisfaction survey will be provided to caregivers which will document how satisfied they were using the intervention, if they believed it helped them, if they would choose to use the intervention again and if they would recommend the intervention.
Clinician Satisfaction Survey | 2 years
  Surgeons will be provided with a self-report survey asking their satisfaction with the technology, the patients' immersion with the technology, and the desire for use in future procedures based on a 1-5 scale.
Cost difference between general anesthesia and virtual reality | 2 years
  Hospital cost data for the procedure will be collected. The difference in cost for patients using general anesthesia versus using virtual reality will then be calculated
Change in Anxiety Scale | 2 years
  Participants will fill out a survey to document their anxiety during and after the procedure. Anxiety will be measured on a visual analogue scale using the Childhood Anxiety Meter (0-10) where participants will fill in a scale of how anxious they were during and after the procedure. Higher values represent a worse outcome (i.e. higher level of anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Chao, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329